CLINICAL TRIAL: NCT02757664
Title: Shock Wave Therapy, Associated to Eccentric Strengthening Versus Isolated Eccentric Strengthening for Treating Insertional Achilles Tendinopathy: Double Blinded Randomized Clinical Trial
Brief Title: Clinical Trial to Evaluate the Adjuvant Effect of Shock Wave Therapy in the Insertional Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Nacime Salomão Barbachan Mansur, Medical Doctor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8094833648737701
Record Dates: First submitted 2016-04-26; First posted 2016-05-02 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Achilles Tendinitis; Tendinopathy
Keywords: achilles; tendinopathy; Physical Therapy Modalities; High-Energy Shock Waves
MeSH Terms: conditions — Tendinopathy | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shock wave plus eccentric exercises (Active Comparator): Shock wave therapy associated with eccentric exercises rehabilitation program.
  Interventions: Device: Shock Wave Therapy; Other: Eccentric Exercises
- Placebo plus eccentric exercises (Placebo Comparator): Placebo associated with eccentric exercises rehabilitation program.
  Interventions: Other: Eccentric Exercises; Device: Placebo

INTERVENTIONS:
Device: Shock Wave Therapy — Appliance of radial shock waves with the BLT600 equipment (BTL Medical Technologies - Canada), the intensity being 2000 to 3000 pulses, 7 to 10Hz of frequency, and 1,5 a 2,5Bar of intensity per application; Appliance on the first day of treatment (D0), repeated on the second week after the first intervention (2nd week) and four weeks after the first intervention (4th week).
  Other Names: radial shock waves
  Arms: Shock wave plus eccentric exercises
Other: Eccentric Exercises — 12 weeks, starting on the same day of the first appliance. The patient will practice the exercises standing on tiptoes and will perform exercises of passive ankle extension (dorsiflexion), three series of 15 repetitions, with the knee stretched, and three series of 15 repetitions with the knee flexed by 20 degrees.
  Other Names: Alfredson eccentric strengthening protocol
Device: Placebo — Placing of the apparatus´ therapeutic head with the support that impedes the shock wave propagation directly on the appliance field; Appliance of radial shock waves with the BLT600 equipment (BTL Medical Technologies - Canada), the intensity being 2000 to 3000 pulses, 7 to 10Hz of frequency, and 1,5 a 2,5Bar of intensity per application; Appliance on the first day of treatment (D0), repeated on the second week after the first intervention (2nd week) and four weeks after the first intervention (4th week).
  Arms: Placebo plus eccentric exercises

SUMMARY:
Background: There is no consensus regarding the treatment of insertional tendinopathies. The good results of the eccentric training in the management of the non-insertional Achilles tendinopathy were not reproducible in the insertional disease. Shock wave therapy is described as an alternative to these patients.

Hypothesis: The shock wave therapy allied to the eccentric strengthening protocol presents better results that the eccentric strengthening associated to placebo.

Design: Double blinded (outcome assessor and patient) randomized clinical trial, with the use of placebo, in parallel groups.

Materials and Methods: Nine-three patients with chronic insertional tendinopathy will be enrolled in a randomized trial. Participants will be divided in two groups, one containing the combination of shock wave and eccentric exercises as treatment and the other comprehending the exercises assembled to placebo. The assessment of outcomes will occur in 2, 4, 6, 12 and 24 weeks of the beginning of the study. Patients will be evaluated for pain, activity and function by the VISA-A (the Victorian Institute of Sport Assessment-Achilles [VISA-A] questionnaire).

DETAILED DESCRIPTION:
Introduction: The insertional tendinopathy occurs in the Achilles attachment to the tuberosity of the calcaneus bone and up to 2 cm proximal to the tuberosity. It is generally associated to a traction enthesophyte (upper spur), to Haglund deformity (pump bump) and to pre and retro achilles bursitis. Nowadays, it is considered that its cause is multi-factorial, comprehending mechanical, vascular, neural and genetic factors. Historically, the disease´s initial treatment is based on motor physiotherapy, via the eccentric strengthening of the tendon. If, on the one hand, the results for non-insertional tendinopathy were encouraging, 82% of them being duly successful, the insertional tendinopathy, on the other hand, produced a rate of improvement ranging between 32 and 67% of the patients, according to the present studies.

The failure of the traditional treatment normally leads the patients to surgery frequently associated to complications, such as wound necrosis and tendon rupture. More recently, the therapy with shock waves is being used in the treatment of pseudo-arthrosis and several types of tendinopathy.

Several studies showed the above mentioned effects of the shock wave therapy may theoretically stimulate neovascularization and of the collagen production that, besides being important in the healing process, also permits several clinical usages, such as the skin healing treatment, the pseudo-arthrosis and several tendinopathies, including the Achilles insertional tendinopathy. The shock wave therapy is being progressively more studied. Recent works have presented good results with the technique however; the evidences are still insufficient to represent a consensus regarding the indication of this treatment.

The objective of the present study is compare the effectiveness of eccentric strengthening protocol with and without shockwave therapy considering the VISA-A.

Hypothesis: The shock wave therapy allied to the eccentric strengthening protocol presents better results that the eccentric strengthening associated to placebo.

Material and Method Design Double blind randomized clinical trial, with the use of placebo, in parallel groups Setting The study will be conducted at Hospital São Paulo - University Hospital of UNIFESP (HSP-UNIFESP), in the Orthopedics and Traumatology Department (DOT) and in CPRT - Centre of Tissue Research and Regeneration (DOT/EPM-UNIFESP); linked to a FINEP project regarding Shock Waves.

Inclusion Criteria: Older than 18 and younger than 65 years of age, both genders; Pain symptoms in the calcaneus tendon insertion region over the last three months; Clinical diagnosis: presence of pain at palpation of the tendinous insertion region in the calcaneus bone (and up to 2cm close to this region) and the occurrence of increase of the region´s volume; Indication of tendinopathy in the Ultra Sound done at the previous health center or by a certified doctor; Lateral X-ray view of the calcaneus, showing any of the associated conditions (Haglund, enthesophyte or intra-substantial calcification).

Exclusion Criteria: Previous surgery involving the affected foot or ankle; History or documented evidence of autoimmune or peripheral vascular diseases; History or documented evidence of peripheral neuropathy (nervous compression syndrome, tarsal tunnel syndrome).History or documented evidence of systemic inflammatory disease a (rheumatoid arthritis, spondylitis, Reiter Syndrome, etc.); Non-Insertional or mixed tendinopathy (insertional and non-insertional); Previous infiltration in the affected tendon over the six months preceding the initial assessment; Beginning of the present pain, due to a trauma; Gross or congenital deformity overweighting the triceps sural muscle, being the main aetiology of the present disease; Pregnancy; Any condition that represents a contraindication of the proposed therapies; Any physical or social limitation that makes the protocol continuation unviable; Impossibility or incapacity to sign the Free Informed Consent Form; History or documented evidence concerning the blood coagulation disorders (treatment with anti-coagulant, excluding aspirin); Use of heart pacemaker;

Sampling: calculation considers a standard deviation of 16.2; the clinical difference to be detected corresponds to 3,3 with sampling error of 5%. It was calculated considering 93 patients divided in two groups in a randomized way. The sampling amount was defined according to the methodology indicated in Attachment I, where, based on the Central Limit Theorem and Laws of Large Numbers, this sampling size guarantees the reliability of the statistics.

Randomization: The randomization sequence will be generated via computing software (http://www.randomizer.org/form.htm), producing a list from 1 - x, and each number will be related to a sole treatment method. Investigators will perform a randomization with interchanged blocks, with the same number of patients in each group.

Allocation: The patients will have to fill out an initial questionnaire in order to be selected (Attachment 1). After that, the assistant doctor will do the physical diagnostic examination of the patient. Then, the US and XRay procedures will take place, in order complete the diagnostic assessment. The patient will be included in the protocol and duly randomized after the diagnostic confirmation is done via anamnesis and physical examination, and also after completion of supplementary tests, signature of the Informed Consent Form, and fulfilment of all the inclusion criteria and non-adequacy to the exclusion criteria. The following data will be collected to do the epidemiological: analysis of the lesions and interventions: Body mass index, Sex, Age, Sports practice (Yes/No), Presence of Haglung Deformity (Y/N), and the Presence of Enthesophyte (Y/N). Each non-transparent sealed envelope, numbered from 1 to 93, will contain either a paper with the word "physiotherapy" or with the words "physiotherapy and shock wave". Each treatment method will have the same number of envelopes. The patients will be initially assessed individually, being randomized and allocated in the same way. The intervention procedures will be the same, with the same positioning and preparations, but differing regarding the existence of a support at the applicator head of the shock wave apparatus in the group of patients without shock wave.

Blinding: Neither the patient nor the evaluator doctor will have access to the protocol test applied to each patient.

The patient will be included in the study after the diagnostic confirmation is done by medical history and physical examination, and also after completion of subsidiary tests (US), signature of the Informed Consent Form, and fulfilment of all the inclusion criteria and non-adequacy to the exclusion criteria.

Intervention: Utilization of shock waves: Appliance of US gel on the region that will receive the shock wave; Appliance of radial shock waves with the BLT600 equipment (BTL Medical Technologies - Canada), the intensity being 2000 to 3000 pulses, 7 to 10Hz of frequency, and 1,5 a 2,5Bar of intensity per application; Appliance on the first day of treatment (D0) as described above, repeated on the second week after the first intervention (2nd week) and four weeks after the first intervention (4th week).

Group without Shock wave: Appliance of US gel on the region that will receive the shock wave; Placing of the apparatus´ therapeutic head with the support that blocks the shock wave propagation directly on the appliance field; Appliance of radial shock waves with the BLT600 equipment (BTL Medical Technologies - Canada), the intensity being 2000 to 3000 pulses, 7 to 10Hz of frequency, and 1,5 a 2,5Bar of intensity per application; Appliance on the first day of treatment (D0) as described above, repeated on the second week after the first intervention (2nd week) and four weeks after the first intervention (4th week).

Eccentric Exercises The groups will be submitted to Alfredson eccentric strengthening protocol for 12 weeks, starting on the same day of the first appliance. The exercises will be shown to the patients by the assistant doctor, and a booklet (Attachment 2) will be handed out, with detailed explanation concerning the protocol to be followed.

Secondary Conclusion: EVA (Visual Analogue Scale); AOFAS; SF-12; Algometry (pain threshold and VAS with 3kg) Follow up: The patients must return to the ambulatory for clinical assessment at 2 weeks, 4 weeks, 6 weeks, 8 weeks, 3 months and 6 months after the beginning of the protocol.

Assessment Scores: The questionnaires VISA-A, EVA, AOFAS and SF-12 will be applied in the first consultation. The patient will be also assessed with the same questionnaires at the intervals of 1, 3 and 6 months of the protocol.

Statistical Analysis: After collecting information we will define the results, with descriptive analysis for the quantitative variables (interval of 95% of reliability for the average/mean). The qualitative variables will require the Comparison of Two Proportions via relative frequency analysis. The Pearson Correlation will be used to check the relation between quantitative variables, and the Chi-Square test will be utilized in relation to qualitative variables. The ANOVA test will be used to compare the two techniques based on their average.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 and younger than 65 years of age, both genders;
* Pain symptoms in the calcaneus tendon insertion region over the last three months;
* Clinical diagnosis: presence of pain at palpation of the tendinous insertion region in the calcaneus bone (and up to 2cm close to this region) and the occurrence of increase of the region´s volume;
* Indication of tendinopathy in the Ultra Sound done at the previous health center or by a certified doctor;
* Lateral X-ray view of the calcaneus, showing any of the associated conditions (Haglund, enthesophyte or intra-substantial calcification).

Exclusion Criteria:

* Previous surgery involving the affected foot or ankle; History or documented evidence of autoimmune or peripheral vascular diseases;
* History or documented evidence of peripheral neuropathy (nervous compression syndrome, tarsal tunnel syndrome).
* History or documented evidence of systemic inflammatory disease a (rheumatoid arthritis, spondylitis, Reiter Syndrome, etc.)
* History or documented evidence of loss of sensibility in the foot or ankle;
* Non-Insertional or mixed tendinopathy (insertional and non-insertional);
* Previous infiltration in the affected tendon over the six months preceding the initial assessment;
* Beginning of the present pain, due to a trauma;
* Gross or congenital deformity overweighting the triceps sural muscle, being the main aetiology of the present disease.
* Pregnancy;
* Any condition that represents a contraindication of the proposed therapies;
* Any physical or social limitation that makes the protocol continuation unviable;
* Impossibility or incapacity to sign the Free Informed Consent Form;
* History or documented evidence concerning the blood coagulation disorders (treatment with anti-coagulant, excluding aspirin);
* Use of heart pacemaker;
* Presence of infectious process (superficial on skin and cellular tissue, or deep in the bone) in the region to be treated;
* Non-palpable anterior or posterior tibial pulse; or abnormal capillary filling;
* Tumour lesions (primary or secondary tumours).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
VISA-A Score change | 0 - 2 weeks - 4 weeks - 6 weeks - 12 weeks - 24 weeks
  Victorian Institute of Sports Assessment - Achilles

SECONDARY OUTCOMES:
VAS - Pain assessment (change) | 0 - 2 weeks - 4 weeks - 6 weeks - 12 weeks - 24 weeks
  Visual Analogue Scale
AOFAS Hindfoot Scale (change) | 0 - 2 weeks - 4 weeks - 6 weeks - 12 weeks - 24 weeks
  American Orthopaedic Foot and Ankle Society Hindfoot Scale
SF-12 (change) | 0 - 2 weeks - 4 weeks - 6 weeks - 12 weeks - 24 weeks
  Short Form (SF-12) Health Survey
Pain threshold at Algometry (change) | 0 - 2 weeks - 4 weeks - 6 weeks - 12 weeks - 24 weeks
  Algometry in the most painful point at the participant's heel
VAS with 3kg of pressure in the Algometer (change) | 0 - 2 weeks - 4 weeks - 6 weeks - 12 weeks - 24 weeks
  Pain assessment by Visual Analogue Scale with 3kg of pressure in the most painful point at the participant's heel

CONTACTS AND LOCATIONS:
Overall Officials: Nacime SB Mansur, MD, Principal Investigator — Researcher; Marcel JS Tamaoki, PhD, Study Director — Researcher
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
According to the ICMJE data sharing police, the datasets supporting the conclusions of this article are available at DataDryard (Mansur, Nacime Salomão Barbachan; Tamaoki, Marcel Jun Sugawara (2020), SHOCK WAVE THERAPY ASSOCIATED WITH ECCENTRIC STRENGTHENING VERSUS ISOLATED ECCENTRIC STRENGTHENING FOR ACHILLES INSERTIONAL TENDINOPATHY TREATMENT: A DOUBLE BLINDED RANDOMIZED CLINICAL TRIAL, Dryad Dataset, https://doi.org/10.5061/dryad.jq2bvq86k) and available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Indefinitely
Access Criteria: Validated researcher

REFERENCES:
- [Background] Den Hartog BD. Insertional Achilles tendinosis: pathogenesis and treatment. Foot Ankle Clin. 2009 Dec;14(4):639-50. doi: 10.1016/j.fcl.2009.08.005. PMID 19857838
- [Background] Irwin TA. Current concepts review: insertional achilles tendinopathy. Foot Ankle Int. 2010 Oct;31(10):933-9. doi: 10.3113/FAI.2010.0933. No abstract available. PMID 20964977
- [Background] Magnan B, Bondi M, Pierantoni S, Samaila E. The pathogenesis of Achilles tendinopathy: a systematic review. Foot Ankle Surg. 2014 Sep;20(3):154-9. doi: 10.1016/j.fas.2014.02.010. Epub 2014 Mar 12. PMID 25103700
- [Background] Wang CJ, Wang FS, Yang KD, Weng LH, Hsu CC, Huang CS, Yang LC. Shock wave therapy induces neovascularization at the tendon-bone junction. A study in rabbits. J Orthop Res. 2003 Nov;21(6):984-9. doi: 10.1016/S0736-0266(03)00104-9. PMID 14554209
- [Background] Hsu RW, Hsu WH, Tai CL, Lee KF. Effect of shock-wave therapy on patellar tendinopathy in a rabbit model. J Orthop Res. 2004 Jan;22(1):221-7. doi: 10.1016/S0736-0266(03)00138-4. PMID 14656684
- [Background] Wang CJ, Huang HY, Pai CH. Shock wave-enhanced neovascularization at the tendon-bone junction: an experiment in dogs. J Foot Ankle Surg. 2002 Jan-Feb;41(1):16-22. doi: 10.1016/s1067-2516(02)80005-9. PMID 11858601
- [Background] Maffulli G, Hemmings S, Maffulli N. Assessment of the Effectiveness of Extracorporeal Shock Wave Therapy (ESWT) For Soft Tissue Injuries (ASSERT): An Online Database Protocol. Transl Med UniSa. 2014 Apr 8;10:46-51. eCollection 2014 Sep. PMID 25147767
- [Background] Mani-Babu S, Morrissey D, Waugh C, Screen H, Barton C. The effectiveness of extracorporeal shock wave therapy in lower limb tendinopathy: a systematic review. Am J Sports Med. 2015 Mar;43(3):752-61. doi: 10.1177/0363546514531911. Epub 2014 May 9. PMID 24817008
- [Background] Speed C. A systematic review of shockwave therapies in soft tissue conditions: focusing on the evidence. Br J Sports Med. 2014 Nov;48(21):1538-42. doi: 10.1136/bjsports-2012-091961. Epub 2013 Aug 5. PMID 23918444
- [Background] Al-Abbad H, Simon JV. The effectiveness of extracorporeal shock wave therapy on chronic achilles tendinopathy: a systematic review. Foot Ankle Int. 2013 Jan;34(1):33-41. doi: 10.1177/1071100712464354. PMID 23386759
- [Background] Notarnicola A, Moretti B. The biological effects of extracorporeal shock wave therapy (eswt) on tendon tissue. Muscles Ligaments Tendons J. 2012 Jun 17;2(1):33-7. Print 2012 Jan. PMID 23738271
- [Background] Wilson M, Stacy J. Shock wave therapy for Achilles tendinopathy. Curr Rev Musculoskelet Med. 2010 Nov 26;4(1):6-10. doi: 10.1007/s12178-010-9067-2. PMID 21475558
- [Background] Rompe JD, Furia J, Maffulli N. Eccentric loading compared with shock wave treatment for chronic insertional achilles tendinopathy. A randomized, controlled trial. J Bone Joint Surg Am. 2008 Jan;90(1):52-61. doi: 10.2106/JBJS.F.01494. PMID 18171957
- [Background] Furia JP. High-energy extracorporeal shock wave therapy as a treatment for chronic noninsertional Achilles tendinopathy. Am J Sports Med. 2008 Mar;36(3):502-8. doi: 10.1177/0363546507309674. Epub 2007 Nov 15. PMID 18006678
- [Background] Rompe JD, Nafe B, Furia JP, Maffulli N. Eccentric loading, shock-wave treatment, or a wait-and-see policy for tendinopathy of the main body of tendo Achillis: a randomized controlled trial. Am J Sports Med. 2007 Mar;35(3):374-83. doi: 10.1177/0363546506295940. Epub 2007 Jan 23. PMID 17244902
- [Background] Furia JP. High-energy extracorporeal shock wave therapy as a treatment for insertional Achilles tendinopathy. Am J Sports Med. 2006 May;34(5):733-40. doi: 10.1177/0363546505281810. PMID 16627628
- [Background] Costa ML, Shepstone L, Donell ST, Thomas TL. Shock wave therapy for chronic Achilles tendon pain: a randomized placebo-controlled trial. Clin Orthop Relat Res. 2005 Nov;440:199-204. doi: 10.1097/01.blo.0000180451.03425.48. PMID 16239807
- [Background] Furia JP. [Extracorporeal shockwave therapy in the treatment of chronic insertional Achilles tendinopathy]. Orthopade. 2005 Jun;34(6):571-8. doi: 10.1007/s00132-005-0806-9. German. PMID 15909176
- [Background] Perlick L, Schiffmann R, Kraft CN, Wallny T, Diedrich O. [Extracorporal shock wave treatment of the achilles tendinitis: Experimental and preliminary clinical results]. Z Orthop Ihre Grenzgeb. 2002 May-Jun;140(3):275-80. doi: 10.1055/s-2002-32475. German. PMID 12085292
- [Background] Wang CJ, Chen HS, Chen CE, Yang KD. Treatment of nonunions of long bone fractures with shock waves. Clin Orthop Relat Res. 2001 Jun;(387):95-101. doi: 10.1097/00003086-200106000-00013. PMID 11400901
- [Background] Wang CJ, Huang HY, Chen HH, Pai CH, Yang KD. Effect of shock wave therapy on acute fractures of the tibia: a study in a dog model. Clin Orthop Relat Res. 2001 Jun;(387):112-8. doi: 10.1097/00003086-200106000-00015. PMID 11400871
- [Background] Meirer R, Kamelger FS, Huemer GM, Wanner S, Piza-Katzer H. Extracorporal shock wave may enhance skin flap survival in an animal model. Br J Plast Surg. 2005 Jan;58(1):53-7. doi: 10.1016/j.bjps.2004.04.027. PMID 15629167
- [Background] Sayana MK, Maffulli N. Eccentric calf muscle training in non-athletic patients with Achilles tendinopathy. J Sci Med Sport. 2007 Feb;10(1):52-8. doi: 10.1016/j.jsams.2006.05.008. Epub 2006 Jul 7. PMID 16828343
- [Background] Fahlstrom M, Jonsson P, Lorentzon R, Alfredson H. Chronic Achilles tendon pain treated with eccentric calf-muscle training. Knee Surg Sports Traumatol Arthrosc. 2003 Sep;11(5):327-33. doi: 10.1007/s00167-003-0418-z. Epub 2003 Aug 26. PMID 12942235
- [Background] Ohberg L, Alfredson H. Effects on neovascularisation behind the good results with eccentric training in chronic mid-portion Achilles tendinosis? Knee Surg Sports Traumatol Arthrosc. 2004 Sep;12(5):465-70. doi: 10.1007/s00167-004-0494-8. Epub 2004 Apr 2. PMID 15060761
- [Result] Kearney R, Costa ML. Insertional achilles tendinopathy management: a systematic review. Foot Ankle Int. 2010 Aug;31(8):689-94. doi: 10.3113/FAI.2010.0689. PMID 20727317
- [Result] Sussmilch-Leitch SP, Collins NJ, Bialocerkowski AE, Warden SJ, Crossley KM. Physical therapies for Achilles tendinopathy: systematic review and meta-analysis. J Foot Ankle Res. 2012 Jul 2;5(1):15. doi: 10.1186/1757-1146-5-15. PMID 22747701
- [Result] Saxena A, Ramdath S Jr, O'Halloran P, Gerdesmeyer L, Gollwitzer H. Extra-corporeal pulsed-activated therapy ("EPAT" sound wave) for Achilles tendinopathy: a prospective study. J Foot Ankle Surg. 2011 May-Jun;50(3):315-9. doi: 10.1053/j.jfas.2011.01.003. Epub 2011 Mar 15. PMID 21406328
- [Result] Hart L. Shock-wave treatment was more effective than eccentric training for chronic insertional achilles tendinopathy. Clin J Sport Med. 2009 Mar;19(2):152-3. doi: 10.1097/01.jsm.0000347357.41069.27. No abstract available. PMID 19451774
- [Result] Rompe JD, Furia J, Maffulli N. Eccentric loading versus eccentric loading plus shock-wave treatment for midportion achilles tendinopathy: a randomized controlled trial. Am J Sports Med. 2009 Mar;37(3):463-70. doi: 10.1177/0363546508326983. Epub 2008 Dec 15. PMID 19088057
- [Result] Rasmussen S, Christensen M, Mathiesen I, Simonson O. Shockwave therapy for chronic Achilles tendinopathy: a double-blind, randomized clinical trial of efficacy. Acta Orthop. 2008 Apr;79(2):249-56. doi: 10.1080/17453670710015058. PMID 18484252
- [Result] Mafi N, Lorentzon R, Alfredson H. Superior short-term results with eccentric calf muscle training compared to concentric training in a randomized prospective multicenter study on patients with chronic Achilles tendinosis. Knee Surg Sports Traumatol Arthrosc. 2001;9(1):42-7. doi: 10.1007/s001670000148. PMID 11269583
- [Derived] Mansur NS, Faloppa F, Belloti JC, Ingham SJ, Matsunaga FT, Santos PR, Santos BS, Carrazzone OL, Peixoto G, Aoyama BT, Tamaoki MJ. Shock wave therapy associated with eccentric strengthening versus isolated eccentric strengthening for Achilles insertional tendinopathy treatment: a double-blinded randomised clinical trial protocol. BMJ Open. 2017 Jan 27;7(1):e013332. doi: 10.1136/bmjopen-2016-013332. PMID 28132005